CLINICAL TRIAL: NCT06285279
Title: Evaluation of the Safety and Efficacy of the BCMA/CD19 Dual Targeted CAR-T Cell in Participants With Autoimmune Kidney Diseases: A Single-center Exploratory Clinical Study
Brief Title: The BCMA/CD19 Dual Targeted CAR-T Cell in Participants With Autoimmune Kidney Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Professor, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-2401
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Lupus Nephritis; ANCA-associated Vasculitis; Membranous Nephropathy - PLA2R Induced; IgG4-Related Diseases
MeSH Terms: conditions — Lupus Nephritis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Administration of the BCMA/CD19 dual targeted CAR-T cells Four dose groups of 0.1×10^6 CAR-T/kg, 0.3×10^6 CAR-T/kg, 1.0×10^6 CAR-T/kg, and 3.0×10^6 CAR-T/kg FKC288 are designed in this study.
  Each dose group plans to enroll 1-2 or 3-6 participants with relapsed or refractory autoimmune-mediated kidney diseases (such as lupus nephritis, ANCA-associated vasculitis, membranous nephropathy, IgG4-related diseases) according to observed DLT.
  the BCMA/CD19 dual targeted CAR-T cells will be intravenously infused at least 24 hours after lymphodepletion preconditioning. According to the assigned dose group, the designated dose of the BCMA/CD19 dual targeted CAR-T cells will be infused in a single infusion within 30 minutes on day 0.
  Interventions: Drug: FKC288

INTERVENTIONS:
Drug: FKC288 — The autologous dual target BCMA/CD19-CAR-T cell of this study is obtained by infecting T cells with anti-BCMA/CD19-CAR lentiviral vectors.
  Administration method: intravenous infusion； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This study is a single-center, open-label, dose-escalation exploratory clinical trial, expected to enroll 6 to 12 participants. It will use a BOIN (Bayesian Optimal Interval) design for dose escalation, with four predetermined dose groups (0.3×10^6 cells/kg, 1.0×10^6 cells/kg, 3.0×10^6 cells/kg, and an alternative dose of 0.1×10^6 cells/kg). Each dose group plans to enroll 1-2 or 3-6 participants with relapsed or refractory autoimmune-mediated kidney diseases (such as lupus nephritis, ANCA-associated vasculitis, membranous nephropathy, and IgG4-related diseases).

DETAILED DESCRIPTION:
A leukapheresis procedure will be performed to manufacture FKC288 chimeric antigen receptor (CAR) modified T cells. Bridging therapy is allowed between PBMC collection and lymphodepletion. Lymphodepletion with fludarabine and cyclophosphamide was performed for three consecutive days. After 1-day rest, subjects will receive a single dose infusion of the BCMA/CD19 dual targeted CAR-T cells at 0.1, 0.3, 1.0, or 3.0x 10^6 CAR+ T cells/Kg. Subjects will be followed in the study for a minimum of 2 years after FKC288 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must personally sign an informed consent form approved by the Ethics Committee before the start of the study.
2. Participants must be aged ≥18 and ≤65 years.
3. Disease-specific inclusion criteria:

   Active, relapsing, refractory Lupus Nephritis (LN):

   LN diagnosed by kidney biopsy within the last 2 years, with pathological types III, IV, or V, and a chronicity index (CI) score≤3

   Meets one of the following criteria:

   Refractory LN, defined as no remission after at least one standard regimen (CTX and/or MMF) for 6 months.

   Relapsing LN, defined as a need to increase steroid dosage to control disease activity during maintenance treatment.

   Clinical criteria: eGFR > 45 ml/min/1.73 m²; urinary protein quantification ≥ 1.5g/24h; SLE-DAI score ≥ 8.

   ANCA-associated vasculitis (AAV) patients:

   Diagnosed as AAV according to the 2012 Chapel Hill Consensus Conference criteria, meeting one of the following:

   Newly diagnosed AAV with renal involvement:

   Renal involvement must meet both:

   Kidney biopsy showing pauci-immune necrotizing glomerulonephritis. Urinary red blood cells >30/high power field.

   Relapsing or refractory AAV:

   Relapse: Defined as an increase in BVAS V3.0 score of ≥1 after remission, requiring adjustment of immunosuppressive treatment to regain remission.

   Refractory: Defined as a) less than 50% reduction in BVAS V3.0 after 6 weeks of standard induction treatment; or b) persistent disease activity (BVAS V3.0 ≥3) after 12 weeks of treatment.

   Membranous nephropathy (MN) patients:

   Tissue biopsy diagnosed as aPLA2R-related membranous nephropathy.

   Clinical criteria for high-risk or relapsing/refractory membranous nephropathy:

   High-risk patients:

   Defined as meeting any of the following: eGFR normal, urinary protein >3.5g/d, ACEI/ARB treatment for 6 months with <50% reduction in urinary protein, combined with serum albumin <25g/l or aPLA2R >50RU/ml; or eGFR <60ml/min/1.73m², and/or urinary protein >8g/d for over 6 months.

   Refractory/relapsing membranous nephropathy patients:

   Refractory: Defined as resistance to previous immunosuppressive treatment (persistent urinary protein ≥3.5g/d with <50% reduction compared to baseline).

   Relapse: Defined as complete or partial remission achieved with previous immunosuppressive treatment, followed by reappearance of urinary protein ≥3.5g/d.

   eGFR ≥ 45 ml/min/1.73 m².

   IgG4-related disease patients:

   Meeting the 2019 ACR/EULAR diagnostic criteria for IgG4-related disease, and meeting one of the following:

   Newly diagnosed active IgG4-related disease (Respond Index (RI) ≥3).

   Refractory or relapsed IgG4-related disease:

   Refractory: Defined as no remission with steroid or steroid plus immunosuppressant treatment (no clinical or imaging improvement, RI decrease <2) Relapse: Defined as new progression or recurrence of clinical symptoms or imaging findings in a patient who had achieved remission, with or without elevated blood IgG4 (RI increase≥2)
4. Expected survival ≥ 12 weeks.
5. ECOG performance status ≤ 2.
6. Female participants of childbearing potential must agree to use effective contraception from the day of signing the informed consent until 365 days after the infusion. Effective contraception is defined as abstinence or the use of a contraceptive method with a failure rate of <1% per year.
7. Participants must have adequate organ function, meeting all of the following criteria before enrollment:

   1. Absolute neutrophil count ≥ 1.0×10⁹/L [Granulocyte colony-stimulating factor (G-CSF) support is allowed, but no supportive treatment should be received within 7 days before the assessment].
   2. Platelet count ≥ 50×10⁹/L [No transfusion support (including component transfusion) or treatments aimed

Exclusion Criteria:

1. Participants who have received the following previous treatments:

   1.1 Participants who have received gene therapy before enrollment. 1.2 Participants who have been injected with live vaccines within 4 weeks prior to enrollment.

   1.3 Participants who have received other investigational drug treatments within 12 weeks before apheresis.
2. Participants with active malignancies within the past 5 years, except for tumors deemed curable and cured, such as basal or squamous cell carcinoma, cervical or breast carcinoma in situ, etc.
3. Participants who are positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) with abnormal peripheral blood HBV DNA tests (defined as HBV DNA quantification above the lower limit of detection or above the normal reference range of the testing center, or qualitative HBV DNA test positive); positive for Hepatitis C virus (HCV) antibodies with positive peripheral blood HCV RNA; positive for Human Immunodeficiency Virus (HIV) antibodies; positive for Cytomegalovirus (CMV) DNA; positive for syphilis test RPR.
4. Participants with uncontrolled active infections (except for < Grade 2 CTCAE urinary reproductive system infections and upper respiratory infections).
5. Participants with severe heart diseases, including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] class ≥ III), severe arrhythmias.
6. Participants with hypertension or diabetes that cannot be controlled with medication.
7. Participants with unresolved toxic reactions from previous treatments to baseline or ≤ Grade 1 (according to NCI-CTCAE v5.0, except for alopecia and clinically insignificant lab abnormalities).
8. Participants who have undergone major surgery within 2 weeks prior to enrollment or plan to have surgery during the waiting period for infusion or within 12 weeks after receiving study treatment (except for planned minor surgeries under local anesthesia).
9. Participants with solid organ transplants.
10. Pregnant or breastfeeding women.
11. Participants with a history of central nervous system diseases (such as cerebral aneurysm, epilepsy, stroke, dementia, psychosis, etc.) or consciousness disorders.
12. Participants with other unstable systemic diseases as judged by the researcher, including but not limited to severe diseases of the liver, kidneys, gastrointestinal tract, or metabolic diseases requiring medication.
13. Participants are known to have life-threatening allergic reactions, hypersensitivity, or intolerance to FKC288 cellular products or their components.
14. Participants judged by the researcher to have bleeding, severe thrombosis, or hereditary/acquired bleeding and severe thrombosis conditions (including hemophilia, coagulation dysfunction, thrombocytopenia, splenomegaly, etc.), or patients currently undergoing thrombolytic or anticoagulant therapy.
15. Participants who have received any B cell-depleting therapy or non-depleting B cell targeted therapy within 6 months.
16. Participants who have received high-dose methylprednisolone treatment (cumulative dose > 1.5g) or cyclophosphamide pulse therapy within a month.
17. Participants judged by the researcher to be unable to discontinue other immunosuppressants one week before apheresis, or those treated with more than 5 mg/day of prednisone (or equivalent dose of other corticosteroids).
18. AAV patients diagnosed with eosinophilic granulomatosis with polyangiitis (formerly Churg-Strauss syndrome) or with active alveolar hemorrhage.
19. Other conditions deemed by the researcher as unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with dose-limiting toxicity | Within 28 days after the BCMA/CD19 dual targeted CAR-T cells injection infusion
  The number of participants with dose limiting toxicity in each dose group and the type of dose limiting toxicity that occurred.
The proportion of subjects with adverse events | Within 24 weeks after the BCMA/CD19 dual targeted CAR-T cells injection infusion
  All adverse events were evaluated according to NCI-CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Proportion of subjects achieving renal response | Within 6 months after the BCMA/CD19 dual targeted CAR-T cells injection infusion
  The proportion of participants who achieve partial remission (PR) or complete remission (CR) of renal.
Duration of response (DoR) of all subjects | Within 2 years after the BCMA/CD19 dual targeted CAR-T cells injection infusion
  The time from FKC288 infusion to the first assessment of CR/PR until the first assessment of disease progression/relapse or death due to the study disease
Progression-free survival (PFS) of all subjects | Within 2 years after the BCMA/CD19 dual targeted CAR-T cells injection infusion
  Time from the first FKC288 infusion to the first assessment of disease progression/relapse or death from any cause.
Overall survival (OS) of all subjects | Within 2 years after the BCMA/CD19 dual targeted CAR-T cells injection infusion
  Time from the first FKC288 infusion to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No